CLINICAL TRIAL: NCT04915482
Title: Efficacy and Safety of TPO-RAs Combined With Anti-CD20 Antibody in the Treatment of Adult Immune Thrombocytopenia With Autoantibodies Failed to First-line Treatment: a Prospective, Open-label, Nonrandomized, Multicenter Clinical Trial
Brief Title: TPO-RAs Combined With Anti-CD20 Antibody in the Treatment of Adult Immune Thrombocytopenia With Autoantibodies
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020034
Record Dates: First submitted 2021-05-25; First posted 2021-06-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-03

CONDITIONS: Immune Thrombocytopenia (ITP); Autoantibodies; Evan Syndrome; Connective Tissue Diseases
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Evans Syndrome; Connective Tissue Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined use of TPO-RAs with low-dose anti-CD20 antibody (Experimental): The starting dose of eltrombopag is 50-75mg once daily. The starting dose of hetrombopag is 5.0-7.5mg once daily. The starting dose of avatrombopag is 20-40mg once daily. Prior to or within 2 weeks after initiation of TPO-RAs therapy, a single dose of Rituximab at 375mg/m2 or divided doses of Rituximab at 100mg once a week for 2-4 weeks, or a single dose of ortuzumab at 1000mg can be administered.. The dosage will be adjusted according to the results of laboratory examinations and patient tolerance.
  Interventions: Drug: Combined use of TPO-RAs with low-dose anti-CD20 antibody
- The best available therapy other than combined use of TPO-RAs with low-dose anti-CD20 antibody (Active Comparator): The best available therapy except for combined use of TPO-RAs with low-dose anti-CD20 antibody includes but not limited to glucocorticoids, intravenous immunoglobulin, recombinant human thrombopoietin, TPO receptor agonists monotherapy, rituximab monotherapy, immunosuppressants, etc., and the researchers will adjust the treatment plan at any time according to the patient's condition.
  Interventions: Drug: The best available therapy

INTERVENTIONS:
Drug: Combined use of TPO-RAs with low-dose anti-CD20 antibody — Experimental: Combined use of TPO-RAs with low-dose anti-CD20 antibody The starting dose of eltrombopag is 50-75mg once daily. The starting dose of hetrombopag is 5.0-7.5mg once daily. The starting dose of avatrombopag is 20-40mg once daily. Prior to or within 2 weeks after initiation of TPO-RAs therapy, a single dose of Rituximab at 375mg/m2 or divided doses of Rituximab at 100mg once a week for 2-4 weeks, or a single dose of ortuzumab at 1000mg can be administered.. The dosage will be adjusted according to the results of laboratory examinations and patient tolerance.
  Arms: Combined use of TPO-RAs with low-dose anti-CD20 antibody
Drug: The best available therapy — The best available therapy except for combined use of TPO-RAs with low-dose anti-CD20 antibody includes but not limited to glucocorticoids, intravenous immunoglobulin, recombinant human thrombopoietin, TPO receptor agonists monotherapy, rituximab monotherapy, immunosuppressants, etc., and the researchers will adjust the treatment plan at any time according to the patient's condition.
  Arms: The best available therapy other than combined use of TPO-RAs with low-dose anti-CD20 antibody

SUMMARY:
This prospective, open-label, nonrandomized, multicenter clinical trial aims at comparing the efficacy and safety of combined use of TPO-RAs with low-dose anti-CD20 monoclonal antibody vs. the best available therapy（BAT）in adult immune thrombocytopenia with autoantibodies failed (due to intolerance or resistance) to first-line treatment.

DETAILED DESCRIPTION:
This is a prospective, open-label, nonrandomized, multicenter clinical trial aiming at comparing the efficacy and safety of combined use of TPO-RAs with low-dose anti-CD20 monoclonal antibody vs. the best available therapy（BAT）in adult immune thrombocytopenia (ITP) with autoantibodies failed (due to intolerance or resistance) to first-line treatment. The subjects include ITP secondary to connective tissue diseases (including but not limited to systemic lupus erythematosus, Sjogren's syndrome and rheumatoid arthritis), primary ITP with positive antinuclear antibody but not up to the diagnostic criteria of connective tissue diseases, primary Evans syndrome, Evans syndrome secondary to connective tissue diseases, and primary ITP with positive Coomb's test but not up to the diagnostic criteria of Evans syndrome.

Adult ITP patients with autoantibodies (18-65 years) will be nonrandomly divided into the following two treatment groups: 1. combined use of TPO-RAs with low-dose anti-CD20 monoclonal antibody. 2. the best available therapy（BAT）other than combined use of TPO-RAs with low-dose anti-CD20 monoclonal antibody.

The current treatment strategies and possible risks of combined use of TPO-RAs with low-dose anti-CD20 monoclonal antibody in the treatment of ITP with autoantibodies will be fully introduced to the patients by the researchers. Then the patients will be divided into one of the two groups according to the patients' will.

ELIGIBILITY:
Inclusion Criteria:

* The patients have provided written informed consent prior to enrollment.
* 18-65 years old.
* Diagnosed as ITP secondary to connective tissue diseases (including but not limited to systemic lupus erythematosus, Sjogren's syndrome and rheumatoid arthritis), primary ITP with positive antinuclear antibody but not up to the diagnostic criteria of connective tissue diseases, primary Evans syndrome, Evans syndrome secondary to connective tissue diseases, and primary ITP with positive Coomb's test but not up to the diagnostic criteria of Evans syndrome.
* Platelet count<30 ×10^9/L at screening.
* Patients who have received at least one first-line treatment of ITP (glucocorticoid and / or intravenous immunoglobulin) in the past, failed (poor efficacy, or failure to maintain efficacy, or relapse), or had contraindications, intolerance, or refusal of first-line treatment.
* Treatment for ITP (including but not limited to glucocorticoids, recombinant human thrombopoietin (rTPO)) must be completed before enrollment, or the dose must be stable or in a phase of reduction within 2 weeks before enrollment. Immunosuppressants (including but not limited to azathioprine, danazol, cyclosporine A, mycophenolate mofetil) must be finished before entering the group, or the dose must be stable or in the reduction period within 3 months before entering the group.
* Effective contraceptive measures will be taken during the clinical trial.

Exclusion Criteria:

* Thrombocytopenia secondary to thyroid disease.
* Patients with any prior history of arterial or venous thrombosis, and with any of the following risk factors: cancer, Factor V Leiden, ATIII deficiency, and antiphospholipid syndrome.
* Those who had received anti-CD20 monoclonal antibody within 6 months or who had previously failed to respond to low-dose anti-CD20 monoclonal antibody.
* Patients who had failed to respond to the previous use of eltrombopag 75 mg once a day, hetrombopag 7.5mg once a day or avatrombopag 40mg once a day for more than 4 weeks.
* Patients who have received splenectomy within one year or have splenectomy plan within one year.
* Patients with lupus encephalopathy or lupus nephritis.
* Patients with cataract.
* Patients with infectious fever (including but not limited to pulmonary infection) within 1 month or with active infection during screening.
* Existing hepatitis B virus, hepatitis C virus replication or HIV infection.
* Patients with agranulocytosis (ANC <1× 10^9/L), or moderate and severe anemia (HGB < 90g/L). For patients with Evans syndrome, patients with HGB< 60g/L will be excluded.
* Severe liver dysfunction (alanine aminotransferase or glutamic oxaloacetic transaminase > 3×ULN), or bilirubin level > 2×ULN except patients with Evans syndrome.
* Patients with severe cardiac or pulmonary dysfunction.
* Severe renal damage (creatinine clearance < 50 ml/min).
* There were surgical planners during the study.
* History of psychiatric disorder.
* Pregnant or lactating women or those planning to be pregnant during the trial.
* Patients with a history of drug/alcohol abuse (within 2 years before the study).
* Patients that have participated in other experimental researches within one month before enrollment.
* Any other circumstances that the investigator considers that the patient is not suitable to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Platelet response | From the start of study treatment (Day 1) up to the end of week 24
  At weeks 4-24, the proportion of subjects with platelet count (PLT) ≥30×10^9/L and at least 2 times the baseline value in 4 out of 6 consecutive tests (at least 1 week interval between each test).

SECONDARY OUTCOMES:
Platelet response | From the start of study treatment (Day 1) up to the end of week 4, 8 and 12
  Proportion of subjects who achieve response (R) within 4, 8 and 12 weeks of treatment.
Platelet response | From the start of study treatment (Day 1) up to the end of week 4, 8 and 12
  Proportion of subjects who achieve complete response (CR) within 4, 8 and 12 weeks of treatment.
Time to platelet response | From the start of study treatment (Day 1) up to the end of week 24
  Time to response is defined as time from the start of treatment to the first time of achieving a platelet count ≥ 30×10^9/ L and at least doubling of the baseline count during the whole 24 weeks.
Duration of platelet response | From the start of study treatment (Day 1) up to the end of week 24
  Total duration of time a participant with a response of R.
Bleeding score | From the start of study treatment (Day 1) up to the end of week 24
  The incidence and grade of bleeding symptoms according to the World Health Organization Bleeding Scale.
ITP-Patient Assessment Questionnaire | From the start of study treatment (Day 1) up to the end of week 24
  In all participants, ITP-Patient Assessment Questionnaire will be used to assess the health related quality of life before and after treatment.
Changes of disease activity index in patients with systemic lupus erythematosus | From the start of study treatment (Day 1) up to the end of week 24
  The proportion of subjects with improvement of disease activity index in patients with systemic lupus erythematosus according to the SLEDAI standard.
The improvement of symptoms | From the start of study treatment (Day 1) up to the end of week 24
  The proportion of subjects with improvement of symptoms including skin symptom, joint pain, dry mouth and dry eyes.
Improvement in immune indexes | From the start of study treatment (Day 1) up to the end of week 24
  The proportion of subjects with improvement immune indexes including antinuclear antibody, extractable nuclear antigens spectrum and Coomb's test.
Discontinuation rate of glucocorticoids | From the start of study treatment (Day 1) up to the end of week 24
  The proportion of subjects with discontinuation use of glucocorticoids.
Hemoglobin response | From the start of study treatment (Day 1) up to the end of week 24
  The proportion of subjects with Evans syndrome who have a hemoglobin level > 110g/L (female) or > 120g/L (male) in the absence of any recent transfusion and without ongoing hemolysis for 2 consecutive weeks (at least 1 week interval).
Hemoglobin response | From the start of study treatment (Day 1) up to the end of week 24
  The proportion of subjects with Evans syndrome who have a hemoglobin level> 100g/L with at least a 20g/L increase from the pretreatment level for 2 consecutive weeks (at least 1 week interval).
functional assessment of chronic illness therapy-fatigue | From the start of study treatment (Day 1) up to the end of week 24
  In all participants, functional assessment of chronic illness therapy-fatigue questionnaire will be used to assess the health related quality of life before and after treatment.

OTHER OUTCOMES:
Incidence of Toxicity | From the start of study treatment (Day 1) up to the end of week 24
  The proportion of subjects with specific pre-defined toxicity, including fever, hypotension, infection, elevated bilirubin, abnormal liver function, cataract and headache, and unpredictable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Rongfeng Fu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China